CLINICAL TRIAL: NCT04145453
Title: Can Including Genotype Information Increase the Effectiveness of Dietary Interventions? Vegetables Intake and Polymorphism TAS2R38 Gene by Healthy Adults
Brief Title: Vegetables Intake and Polymorphism TAS2R38 Gene by Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UKB 872/19
Record Dates: First submitted 2019-10-03; First posted 2019-10-30 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Healthy Lifestyle; Taste Disorders; Diet Habit
Keywords: TAS2R38 Polymorphism; bitter; taste; PAV; AVI; vegetables; personalized nutrition; genotype; intake; fruit and vegetables
MeSH Terms: conditions — Taste Disorders; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: To achieve the goals of the study, a group of healthy adults will be qualified. Genotype will be assed at the baseline. Consumption of fruit and vegetables will be assessed before and after intervention. The duration of the study will be 20 weeks. Blood results and body analyze will be assessed at the beginning and after the intervention. Overall food consumption will be assessed at the beginning. For the basic characteristics of study participants, their anthropometric and biochemical parameters will be analyzed twice at the baseline and after intervention. The intervention effect, including the TAS2R38 polymorphism, will be analyzed by statistical analysis.
  In a randomized manner volunteers will be assigned to one of three groups: intervention and two control group.
Who Masked: Investigator
Masking Description: lnvestigator is responsible for collecting the questionnaires and anonymizing the data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention group (Experimental): Participants with PAV haplotype will receive personalised dietary recommendations regarding consumption of fruit and vegetables. The information about genotype will be given at the beginning of study.
  Interventions: Behavioral: Intervention genotype personalized nutritional recommendations
- control group 1 (Sham Comparator): Participants with PAV haplotype will receive personalised dietary recommendations regarding consumption of fruit and vegetables, but the information about genotype will be given at the end of study.
  Interventions: Behavioral: Control Group 1 personalized nutritional recommendations
- Control group 2 (Active Comparator): Participants with AVI haplotype will receive general recommendations regarding consumption of fruit and vegetables.
  Interventions: Behavioral: Control Group 2 general nutritional recommendations

INTERVENTIONS:
Behavioral: Intervention genotype personalized nutritional recommendations — Participants will receive personalized nutritional recommendations to increase fruit and vegetables consumption. Information about genotype will be given at the beginning of study
  Other Names: with PAV haplotype
  Arms: intervention group
Behavioral: Control Group 1 personalized nutritional recommendations — Participants will receive genotype personalized nutritional recommendations to increase fruit and vegetables consumption. Information about genotype will be given at the end of study
  Other Names: with PAV haplotype
  Arms: control group 1
Behavioral: Control Group 2 general nutritional recommendations — Participants will receive general nutritional recommendations to increase fruit and vegetables consumption
  Other Names: with AVI haplotype
  Arms: Control group 2

SUMMARY:
Personalized nutrition is one of the most up to date trends in human nutrition and gains much interest of general public and scientists as well. Although we have gained some knowledge on gene-trait associations, the real effectiveness and usefulness of genotype-based nutritional recommendations is unknown. Many personalized nutrition companies are on the market today, some of them use personalized nutrition based on genotype analysis. For this reason, scientific basis of this approach should be clarified.

Our project can thus increase knowledge which can be applied in dietary counseling practice. Although we focus on increase vegetable and fruits intake, the study is designed as a proof of concept.

DETAILED DESCRIPTION:
In humans, the TAS2R38 receptor gene is responsible for differences in the perception of bitter taste. This gene codes for a G protein that is associated with a flavor receptor regulated by phenylthiocarbamide (PTC) and propylthiouracil (PROP) ligands, which by binding to the receptor determines the degree of bitter taste. Cruciferous vegetables contain glucosinolates and isothiocyanates, which resemble PTC and PROP and thereby affect their perception of bitter taste through the TAS2R38 regulated receptor.

The polymorphism of this gene allows to distinguish three phenotypes:

* insensitive to bitter taste [bitter-non tasters]
* moderately sensitive to bitter taste [intermediate-bitter tasters]
* sensitive to bitter taste [bitter taster] Previous studies have shown that people who are carriers of one PAV haplotype experience a bitter taste more than AVI / AVI homozygotes, which are less sensitive to bitter taste. Hence, the TAS2R38 gene polymorphism is associated with nutritional decisions, including choice of vegetables and coffee.

Aim of the study is to verify effectiveness of the genotype based dietary intervention in people with or without polymorphism of TAS2R38 gene.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* injuries, chronic diseases (e.g. diabetes, metabolic syndrome, cancer, hyperthyroidism), recent diet, pregnancy, breastfeeding, limited communication to the extent that no nutritional history can be carried out, eating disorders (according to nutritional history)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Vegetables intake | Baseline, 20 weeks
  Change in frequency of vegatables intake within the group and between the groups; Block vegetables intake screener
TAS2R38 polymorphism | baseline
  genotyping of polymorphism TAS2R38 gene (rsr713598, rs1726866, and rs10246939)

SECONDARY OUTCOMES:
Body Mass (BM) | Baseline, 20 weeks
  change in body mass (kg) within the group and between the groups
Fat free mass (FFM) | Baseline, 20 weeks
  change in FFM (kg) within the group and between the groups
Fat Mass (FM) % | Baseline, 20 weeks
  change in Fat Mass % within the group and between the groups
Waist circumference (WC) | Baseline, 20 weeks
  Change in WC (cm) within the group and between the groups
Total Cholesterol (TChol) | Baseline, 20 weeks
  Changes in TChol (mg/dl) within the group and between the groups
LDL Cholesterol(LDL-Chol) | Baseline, 20 weeks
  Changes in LDL-Chol (mg/dl) within the group and between the groups
HDL Cholesterol (HDL-Chol) | Baseline, 20 weeks
  Changes in HDL-Chol (mg/dl) within the group and between the groups
Triglycerides (TG) | Baseline, 20 week
  Changes in TG (mg/dl) within groups and between groups
Glucose (GLU) | Baseline, 20 weeks
  Changes in GLU (mg/dl) within the group and between the groups
Insulin (INS) | Baseline, 20 weeks
  Changes in INS (ulU/ml) within the group and between the groups
Alanine transaminase (ALAT) | Baseline, 20 weeks
  Changes in ALAT (U/l) within the group and between the groups
aspartate aminotransferase (ASPAT) | Baseline, 20 weeks
  Changes in ASPAT (U/l) within the group and between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Bulczak, Msc, Principal Investigator — Poznan University of Life Science
Locations (1):
- Poznan University of Life Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No